CLINICAL TRIAL: NCT00482430
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled, 2-Period, Cross-Over Clinical Trial to Study the Safety and Efficacy of MK0557 for the Treatment of Cognitive Impairment in Patients With Schizophrenia
Brief Title: MK0557 for the Treatment of Cognitive Impairment in Patients With Schizophrenia (0557-027)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0557-027; MK0557-027; 2007_520
Record Dates: First submitted 2007-05-31; First posted 2007-06-05 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Paranoid Schizophrenia; Schizophrenia
Keywords: Undifferentiated schizophrenia; Residual schizophrenia
MeSH Terms: conditions — Schizophrenia, Paranoid; Schizophrenia | interventions — spiro(cyclohexane-1,3'(1'H)-furo(3,4-C)pyridine)-4-carboxamide, N-(1-(2-fluorophenyl)-1h-pyrazol-3-yl)-1'-oxo-, trans-

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Other): MK0557 10mg tablet qd, crossing over to MK0557 Pbo tablet qd.
  Interventions: Drug: MK0557; Drug: Comparator: Placebo (unspecified)
- 2 (Other): MK0557 Pbo tablet qd, crossing over to MK0557 10mg tablet qd.
  Interventions: Drug: MK0557; Drug: Comparator: Placebo (unspecified)

INTERVENTIONS:
Drug: MK0557 — MK0557 10mg tablet qd for a 15-wk treatment period
Drug: Comparator: Placebo (unspecified) — MK0557 Pbo tablet qd for a 15-wk treatment period

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of an investigational drug for the treatment of cognitive impairment in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patient is clinically stable, on current antipsychotic medication for at least 3 months and current dose for 2 months
* Patient has a 6th grade reading level or better and has completed at least 6 years of formal education
* Females are not pregnant, and those who can have children agree to remain abstinent or use acceptable birth control throughout study
* Patient has had a stable living arrangement for at least 3 months prior to study start
* Patient is in general good health based on screening assessments

Exclusion Criteria:

* Patient has a major disease/disorder that may interfere with cognitive testing (such as mental retardation) and/or pose a risk upon study participation
* Patient has a history of head trauma with loss of consciousness greater than 15 minutes
* Patient has had warfarin treatment, MAO inhibitors, clonazepam, clozapine or St. John's wort within 1 month of screening
* Patient has had ECT treatment within 6 months of screening
* Patient requires treatment with antihistamines or certain other medications listed in the protocol
* Patient has a history of liver disease that has been active within the last 2 years, or a history of cancer within past 5 years
* Patient has a history of alcohol or drug dependence within past year or alcohol or drug abuse within 3 months of screening

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline at 4 weeks of treatment on a sequence of cognitive tests and that MK0557 generally well tolerated | at 4 weeks of treatment

SECONDARY OUTCOMES:
Mean change from baseline at 4 weeks of treatment on neuropsychological tests for executive functioning, episodic memory and working memory | at 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC